CLINICAL TRIAL: NCT01462656
Title: A Post Marketing Surveillance Study to Monitor the Risk of Urinary Retention in Retigabine Users
Brief Title: Risk of Urinary Retention With Retigabine
Status: Terminated | Type: Observational
Why Stopped: This study was halted as the preliminary analysis revealed that the numbers were too low to warrant continuing the project
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115981; WEUKSTV4551 (Other: GSK); EPI40621 (Other: GSK)
Record Dates: First submitted 2011-07-21; First posted 2011-10-31 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Epilepsy
Keywords: anti-epileptic drug; ezogabine; AED polytherapy; epilepsy; AED monotherapy; retigabine; urinary retention
MeSH Terms: conditions — Epilepsy; Urinary Retention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with urinary retention: Patients with urinary retention
  Interventions: Drug: Non-EZG containing AED polytherapy; Drug: EZG containing AED polytherapy; Drug: Non-EZG AED monotherapy; Drug: EZG AED monotherapy

INTERVENTIONS:
Drug: Non-EZG containing AED polytherapy — AED polytherapy without EZG
Drug: EZG containing AED polytherapy — AED polytherapy including EZG
Drug: Non-EZG AED monotherapy — AED monotherapy without EZG
Drug: EZG AED monotherapy — Any off-label use of EZG as monotherapy

SUMMARY:
A prospective cohort study of antiepileptic drug (AED) polytherapy-treated epilepsy patients within the HealthCore Integrated Research Database (HIRD) will be conducted. Following the launch of Ezogabine (EZG), patients initiating a new AED polytherapy regimen will be followed until the earliest of an episode of urinary retention (UR), change in their AED regimen, end of follow-up, or end of study (when the specified sample size of EZG AED polytherapy users has been attained). After the end of study, the incidence of UR during exposures to EZG and non-EZG AED polytherapies will be compared. Polytherapy will be defined as treatment regimen containing at least two different AEDs.

A prospective cohort study of patients who receive EZG under circumstances not indicated in the product label within the HIRD will also be conducted. Following the launch of EZG, epilepsy patients initiating AED monotherapy with EZG as well as non-epilepsy patients initiating EZG for another disease will be followed until the earliest of an episode of UR, change in their AED regimen (if applicable), end of follow-up, or end of study. The incidence of UR during exposure to EZG under circumstances not indicated in the product label will be described. A descriptive analysis of the patients will also be included.

To meet the other secondary objective, non-EZG AED monotherapy users will be identified in the prospective cohort and incidence of UR will be calculated to determine if there is a difference in UR risk between monotherapy and polytherapy AED use.

DETAILED DESCRIPTION:
Epilepsy is one of the most common neurological disorders, with a prevalence of active disease between 0.3 and 1.8% based on population-based studies across the world (0.7% in US) using medical record reviews. These studies have estimated approximately 1.4 million current epilepsy patients in the US alone. Effective seizure control often requires long-term exposure and compliance to various AEDs. Despite the advent of many new AEDs over the past 15 years, approximately 30% of epilepsy patients continue to experience recurrent seizures due to lack of treatment efficacy and discontinuation of therapy due to undesirable side effects or poor treatment compliance. Therefore, an unmet need remains for treatments that can reduce seizure frequency and severity as well as improvements in AED tolerability and safety.

In January 2010, the FDA accepted the new drug application (NDA) for EZG for adjunctive treatment of epilepsy in adults with partial-onset seizures. US market entry is anticipated by 2011. EZG is the first potassium channel opener to reach late stage clinical development for the treatment of epilepsy. EZG's anticonvulsant properties are primarily mediated by opening or activating neuronal voltage-gated potassium channels. The efficacy and safety of EZG as part of polytherapy AED regimens in adults with refractory partial-onset seizures has been demonstrated in one Phase II and two Phase III double-blind, placebo-controlled trials: RESTORE 1 and 2.

In the Phase II study, 399 patients were randomized to four treatment arms (placebo, 600, 900, and 1200 mg/day EZG). The median change from baseline seizure frequency was 13.1% for the placebo group; in comparison, the median change was 23.4% for 600 mg/day, 29.3% for 900 mg/day (p=0.0387), and 35.2% for 1200 mg/day (p=0.0024). RESTORE 1 was conducted in the US and had two arms (placebo and 1200 mg/day EZG), while RESTORE 2 was conducted mainly in Europe and Australia with three different arms (placebo, 600, and 900 mg/day EZG). In RESTORE 1 (n=301), the median reduction in seizure frequency among patients using 1200 mg/day EZG (n=151) was 44% compared with 18% among placebo users (n=150; p<0.001). In RESTORE 2, a significant reduction in partial seizure frequency was found in both EZG doses vs. placebo (p<0.001): 28% for 600 mg/day, 40% for 900 mg/day, and 16% for placebo.During these trials EZG was generally well tolerated; most adverse events (AEs) were mild or moderate with central nervous system (CNS) related AEs (dizziness, somnolence and fatigue) being most common. However, among non-CNS events, an increased incidence of bladder-related AEs, including UR, relative to placebo was observed with EZG, primarily with 1200 mg/day. Among the patients in EZG arms from all trials (n=813), 0.9% experienced UR compared with 0.5% in the placebo arms (n=427). In addition 5% of patients in the EZG arms compared with 3% of patients in the placebo arms experienced urinary symptoms, including dysuria, urinary hesitancy, and UR.

There are concerns that these AEs may reflect the inhibition of bladder contractility secondary to EZG's effects on KCNQ (Kv7) voltage-gated potassium channels in the detrusor muscle of the bladder. However, the limited number of patients exposed to EZG during trials suggests that the risk of UR associated with exposure to EZG has to date been poorly quantified.

A post-marketing safety surveillance study using a US health insurance claims database coupled with medical records review will be implemented to determine the risk of UR associated with exposure to AED polytherapy regimens containing EZG in a real-world setting. The risk of UR among epilepsy patients treated with EZG AED polytherapy will be compared to the risk among epilepsy patients treated with non-EZG AED polytherapy. In addition, both EZG and non-EZG AED polytherapy users will be described in terms of their demographic characteristics, concomitant AED use, co-morbidities, use of medications potentially associated with UR, and medical conditions pre-disposing to UR. Secondarily, off-label usage of EZG will be monitored and described. In addition, the risk of UR among epilepsy patients treated with non-EZG AED monotherapy will be determined.

The primary objective of the study is to quantify the risk of UR associated with exposure to EZG AED polytherapy in a real-world setting. Specific aims include the following:1) to describe patients receiving EZG and non-EZG AED polytherapy in terms of demographics, concomitant AED use, co-morbidities/past medical history, use of medications potentially associated with UR, and medical conditions associated with UR; 2) to determine the magnitude of the risk and time to onset of UR associated with post-marketing use of EZG AED polytherapy, and to determine the incremental risk compared with non-EZG AED polytherapy use; and 3) to determine whether the risk and time to onset of UR associated with non-EZG monotherapy use.

ELIGIBILITY:
Inclusion Criteria:

* Prospective Cohort (indicated use)

  * Patients with at least one medical claim carrying an ICD-9 code for epilepsy. The following ICD-9 codes will be used to identify patients with epilepsy:

    * 345 Epilepsy and recurrent seizures
    * 780.3 Convulsions
    * 780.39 Other convulsions
  * Patients initiating a new AED monotherapy* or polytherapy** following the launch of EZG.
  * At least 6 months of continuous healthcare plan enrolment before initiation of the new AED (monotherapy or polytherapy) following the launch of EZG. This will allow an assessment of baseline co-morbidities and concomitant medication use.
  * Aged ≥18 years at initiation of the new AED (monotherapy or polytherapy).
* Prospective Cohort (non-indicated use)

  * Epilepsy patients initiating EZG AED monotherapy
  * Patients <18 years old initiating EZG for epilepsy
  * Patients initiating EZG for any reason other than epilepsy
  * Patients initiating EZG AED polytherapy with less than six months of continuous healthcare enrolment who were excluded from the cohort described under the primary objective
* Retrospective Cohort

  * Patients with at least one medical claim carrying an ICD-9 code for epilepsy in the three year period preceding the launch of EZG. The following ICD-9 codes will be used to identify patients with epilepsy:

    * 345 Epilepsy and recurrent seizures
    * 780.3 Convulsions
    * 780.39 Other convulsions
  * Patients initiating a new AED monotherapy* or polytherapy** regimen in the three year period preceding the launch of EZG.
  * At least 6 months of continuous healthcare plan enrolment before initiation of the new AED regimen (monotherapy or polytherapy) during the three year period preceding the launch of EZG. This will allow an assessment of baseline co-morbidities and concomitant medication use.
  * Aged ≥18 years at initiation of the new AED (monotherapy or polytherapy).

    * This will include patients substituting an AED monotherapy. **This will include patients switching from a monotherapy to polytherapy regimen and those substituting an AED within an existing polytherapy regimen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study cohorts of interest will be identified from the HealthCore Integrated Research Database (HIRD). The HIRD contains fully adjudicated paid claims from the largest commercially insured population in the US, with dates of service for all non-capitated ambulatory, emergency department, inpatient, and outpatient encounters (including administrative claims for laboratory tests) for members with eligibility at the time of service.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2011-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The risk and time to onset of UR associated with post-marketing use of EZG AED polytherapy, and the incremental risk compared with non-EZG AED polytherapy use. | From initiation of a new AED polytherapy regimen, until the earliest of an episode of UR, change in their AED regimen, end of follow-up, or end of study, whichever comes first, assesed up to three years.

SECONDARY OUTCOMES:
The risk and time to onset of UR among patients using EZG vs. non-EZG AED polytherapy | From initiation of a new AED polytherapy regimen, until the earliest of an episode of UR, change in their AED regimen, end of follow-up, or end of study, whichever comes first, assesed up to three years.
The risk of UR associated with post-marketing use of EZG under circumstances not indicated in the product label | From initiation of a new AED polytherapy regimen, until the earliest of an episode of UR, change in their AED regimen, end of follow-up, or end of study, whichever comes first, assesed up to three years.
The risk of UR among non-EZG AED monotherapy patients and the differential risk in UR for monotherapy versus polytherapy-treated patients | From initiation of a new AED monotherapy regimen, until the earliest of an episode of UR, change in their AED regimen, end of follow-up, or end of study, whichever comes first, assesed up to three years.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline